CLINICAL TRIAL: NCT01041794
Title: Tissue Partitioning in Early Childhood: A Critical Period for Obesity Risk?
Brief Title: Tissue Partitioning in Early Childhood
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Krista Casazza, Krista R. Casazza PhD, RD/Assistant Professor, UAB, University of Alabama at Birmingham
Other Study IDs: F091006004
Record Dates: First submitted 2009-12-30; First posted 2010-01-01 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Changes in Bone Mineral Content; Changes in Bone Marrow Adipose Tissue
Keywords: body composition; fat distribution; exercise; diet
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Samples will be labeled with the study protocol number, a unique identifier, and the date of collection.
  Blood specimens will be obtained by the nursing staff at the PCIR. The PCIR processing lab will process the samples, which will then be stored in a locked freezer at -80oC in the restricted access CNRU Metabolism Core lab (WEBB 337).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
Early childhood (~4-6 years of age) is an important window for determining body composition trajectory and may be a critical period for the development of tissue partitioning patterns that influence later disease risk, including obesity and type 2 diabetes. As adiposity accelerates during this critical period, deposition/ preservation of fat stores may be sustained at the 'expense' of other tissues; i.e. energy homeostasis may be inherently biased toward fat gain. The type and amount of tissue mass accrued in early childhood has implications for metabolic profile, glucose/insulin homeostasis, hormone profile and resting energy expenditure.

The interplay between fat and bone deposition represents a physiologic trait enabling the body to choose between shuttling 'energy' towards accrual of a particular tissue. Plausibly the phenotype underlying obesity and diabetes risk may be determined by the differentiation of cell type (adipocyte, osteocyte, etc.) during this early stage of growth and development. In vitro studies demonstrate transdifferentiation under the influence of specific external stimuli, which can switch phenotypes toward other cell lineages. Further, rodent models have demonstrated that exposure to stimuli (exercise) early in life may prevent excess fat mass accrual in adulthood, even when the stimulus is later removed (animals are no longer exercising). Children's early experiences (engagement in physical activity) may 'environmentally induce' alterations in body composition and predispose individuals to diabetes throughout life (Figure 1).

Hypotheses and Specific Aims: Early growth patterns and cell differentiation may induce long term effects on body composition by impacting biological and hormonal axes that regulate childhood body composition. Body composition comprises not only absolute mass, but also aspects of size, shape and location. To that end, the following specific aims will be evaluated:

1. Quantify body composition, adipose tissue distribution, and relative tissue ratios using magnetic resonance imaging (MRI) and dual-energy x-ray absorptiometry (DXA).

   1. Hypothesis: Early partitioning of 'resources' toward fat mass accrual will lead to decreased gains in bone mass that may persist long-term.
   2. Hypothesis: Partitioning of tissue toward fat at the expense of bone mass (and indirectly, lean mass) will result in adverse effects on glucose/insulin metabolism, total energy expenditure, resting metabolic rate and hormone signaling.
   3. Hypothesis: Children with greater levels of physical activity (energy expenditure) will have greater partitioning towards bone (and lean) mass.
2. Quantify adipose tissue distribution and adipocyte cell size and number using MRI and histological techniques.

   1. Hypothesis: A relatively greater amount of bone marrow adipose tissue will be apparent in those children with low levels of physical activity, resulting in the preferential differentiation of pluripotent stem cells towards adipocytes vs osteocytes in the bone marrow cavity.
   2. A relatively greater adipocyte cell number will be apparent in those children with low levels of physical activity indicating greater differentiation of MSC towards adipocytes vs osteocytes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Aged 3-7 years
* Not taking medications known to affect body composition or metabolism

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children aged three to seven years
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate if early life experiences may induce long term effects on body composition by impacting biological and hormonal axes that regulate childhood body composition. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States